CLINICAL TRIAL: NCT00630942
Title: Open Label Pilot Study Evaluating Minocycline in Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: Minocycline in Primary Sclerosing Cholangitis (PSC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Keith D. Lindor, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 1559-02
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm, active treatment (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 100 mg capsules twice a day before breakfast and before dinner.

SUMMARY:
The purpose of the study is to see how safe and effective minocycline is in the treatment of Primary Sclerosing Cholangitis (PSC).

DETAILED DESCRIPTION:
The purpose of the study is to determine the safety profile of minocycline in patients with PSC and to compare the effects of minocycline on the baseline values of the following parameters: symptoms of pruritus and fatigue, liver biochemistries, Mayo Risk Score, the development of clinical progression and complications of liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Females of childbearing age must have negative pregnancy test within 48 hours of participation and agreement to practice contraception for the duration of the study.
* Age 18 years old and < than 75 years old.
* History of chronic cholestatic disease of at least 6 months duration.
* Serum alkaline phosphatase level at least 1.5 times the upper limit of normal.
* Cholangiography demonstrating intrahepatic and/or extrahepatic biliary obstruction, beading, or narrowing consistent with PSC.
* Liver biopsy consistent with the diagnosis of PSC.
* Patient's informed consent for study participation.

Exclusion Criteria:

* Treatment with tetracyclines, ursodeoxycholic acid, corticosteroids, colchicine, methotrexate, azathioprine, cyclosporine, chlorambucil, budesonide, pentoxifylline, pirfenidone, nicotine, tacrolimus, silymarin, vitamin E or prednisone in the preceding three months.
* Findings highly suggestive of hepatobiliary disease of other etiology complicating PSC.
* Anticipated need for liver transplantation in one year determined by the Mayo model with an estimate of <75% one year survival without transplantation.
* Recurrent variceal bleeding, presence of ascites, or encephalopathy.
* Active drug or alcohol use.
* Pregnancy.
* Breast-feeding.
* Serum creatinine over 1.5 mg/dl.
* Prior history of allergic reactions to antibiotics belonging to the tetracycline family.
* Any condition that, in the opinion of the investigator, would interfere with the patient's ability to complete the study safely or successfully.
* Patients with active inflammatory bowel disease (IBD) requiring specific treatment in the preceding three months, except for maintenance therapy with 5-ASA compounds, or those individuals who have been involved in a trial evaluating any experimental drug for the treatment of IBD in the preceding three months.
* Recurrent ascending cholangitis requiring hospitalization in the past year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and estimate the efficacy at the maximally tolerated dose, 100 mg BID, in 30 patients with PSC. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keith D. Lindor, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States